CLINICAL TRIAL: NCT03615274
Title: Executive Function Training in Childhood Obesity: Food Choice, Quality of Life and Brain Connectivity
Acronym: TOuCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Collaborators: Fundació La Marató de TV3 (Other)
Responsible Party: Principal Investigator, María Ángeles Jurado Luque, Full professor, University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016-16-10
Record Dates: First submitted 2018-07-18; First posted 2018-08-03 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Obesity
Keywords: childhood obesity; cognitive training; executive function; quality of life; neuroimaging; magnetic resonance; connectivity; decision making
MeSH Terms: conditions — Obesity; Pediatric Obesity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Children in the training group must complete home-based executive function training by iPad. At the same time, they are asked to learn basic psychoeducational contents and send pictures of their daily meals. Furthermore, physical activity and sleep patterns are registered over the training period.
  Interventions: Device: Executive function training; Other: Psychoeducation
- Placebo non-adaptive training (Active Comparator): Children in the control group must complete cognitive control tasks. They are also asked to learn basic psychoeducational contents and send pictures of their daily meals. Furthermore, physical activity and sleep patterns are registered over the training period.
  Interventions: Other: Psychoeducation; Device: Placebo non-adaptive training

INTERVENTIONS:
Device: Executive function training — Home-based executive function training with adaptive difficulty, through Cogmed and Cognifit systems over 6 weeks (30-45 minuts/day, 5 days per week). Cognitive training will consist on working memory training (Cogmed, www.cogmed.com) and executive/inhibitory function training (Cognifit, www.cognifit.com).
  Arms: Experimental
Other: Psychoeducation — Learning basic healthy habits through daily Prezi presentations that include healthy food recommendations, funny receipts to families, ideas for exercising, emotion and behavioral management strategies, etc.
Device: Placebo non-adaptive training — Executive function training with non-adaptive difficulty through Cognifit system over 6 weeks (30-45 minuts/day, 5 days per week). Exercices will be the same as the ones in the experimental group but minimizing the executive/working memory component and without incresing difficulty.
  Arms: Placebo non-adaptive training

SUMMARY:
This study evaluates if executive function training in obese children can improve food-related choices and produce cognitive and neuroimaging changes, but also improve psychological and physical status and quality of life measures.

DETAILED DESCRIPTION:
Based on the limited success of current behavioural weight-loss programmes and coupled with data on executive function deficiencies in obesity, this study aims to explore the impact of executive function training on food-related choices, cognitive and neuroimaging outcomes, but also on the psychological and physical status and quality of life measures.

The specific hypotheses are:

1. Obese children undergoing the training programme will perform better than those receiving the control programme in cognitive, emotional state, physical activity and quality of life measures at the end of the intervention and follow-up at 12 months.
2. Obese children receiving the training programme will take better food-related decisions at the end of the intervention and follow-up at 12 months.
3. Obese children receiving the training programme will show changes in brain connectivity, which will be observable immediately at the end of the intervention and during the follow up period at 12 months.
4. There will be an association between changes in neuroimaging biomarkers and food choice, cognitive, emotional, physical and quality of life outcomes in individuals receiving training.

ELIGIBILITY:
Inclusion Criteria:

* Being obese according to the criteria by Cole et al., (2000)

Exclusion Criteria:

* Neurological, psychiatric or developmental disorder.

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2021-01-27 (Actual); Study Completion 2021-01-27 (Actual)

PRIMARY OUTCOMES:
Change from baseline estimated verbal intelligence quotient (IQ) at 12 months | Baseline (T0; 1 week before intervention); follow-up (T2; 12 months after intervention finished)
  Vocabulary subtest (Wechsler intelligence scale for children - Fifth edition, WISC-V). 29 items. Each item is scored 0 or 1 (0=incorrect; 1=correct), yielding a total between 0 and 54.
Change from baseline estimated visuospatial intelligence quotient (IQ) at 12 months | Baseline (T0; 1 week before intervention); follow-up (T2; 12 months after intervention finished)
  Matrix Reasoning subtest (WISC- V). 32 items. Each item is scored 0 or 1 (0=incorrect; 1=correct), yielding a total between 0 and 32.
Change from baseline immediate verbal attention at 8 weeks and at 12 months | Baseline (T0; 1 week before intervention); postraining (T1; 1 week after intervention); follow-up (T2; 12 months after intervention finished)
  Forward Digit Span (WISC-V). 9 items. Each item is scored 0 or 1 (0=incorrect; 1=correct), yielding a total between 0 and 18.
Change from baseline immediate visuospatial attention at 8 weeks and at 12 months | Baseline (T0; 1 week before intervention); postraining (T1; 1 week after intervention); follow-up (T2; 12 months after intervention finished)
  Forward Spatial Span (Wechsler Nonverbal Scale of Ability; WNV). 8 items. Each item is scored 0 or 1 (0=incorrect; 1=correct), yielding a total between 0 and 16.
Change from baseline speed and selective verbal attention at 8 weeks and at 12 months | Baseline (T0; 1 week before intervention); postraining (T1; 1 week after intervention); follow-up (T2; 12 months after intervention finished)
  Reading and counting (Five Digits Test). Total expended time.
Change from baseline speed and selective visual attention at 8 weeks and at 12 months | Baseline (T0; 1 week before intervention); postraining (T1; 1 week after intervention); follow-up (T2; 12 months after intervention finished)
  Children Color Trail Test - I. Total expended time.
Change from baseline sustained visual attention at 8 weeks and at 12 months | Baseline (T0; 1 week before intervention); postraining (T1; 1 week after intervention); follow-up (T2; 12 months after intervention finished)
  Continuous Performance Test -III. Detectability: number of correct responses to non-targets (i.e., the letter X) and to targets (i.e., all other letters). Omissions: number of failures to respond to targets. Comissions: number of incorrect responses to non-targets. Perseverations: number of random or anticipatory responses.
Change from baseline verbal digit working memory at 8 weeks and at 12 months | Baseline (T0; 1 week before intervention); postraining (T1; 1 week after intervention); follow-up (T2; 12 months after intervention finished)
  Backward Digit Span (WISC-V). 9 items. Each item is scored 0 or 1 (0=incorrect; 1=correct), yielding a total between 0 and 18.
Change from baseline visuospatial working memory at 8 weeks and at 12 months | Baseline (T0; 1 week before intervention); postraining (T1; 1 week after intervention); follow-up (T2; 12 months after intervention finished)
  Backward Spatial Span (WNV). 8 items. Each item is scored 0 or 1 (0=incorrect; 1=correct), yielding a total between 0 and 16.
Change from baseline verbal working memory at 8 weeks and at 12 months | Baseline (T0; 1 week before intervention); postraining (T1; 1 week after intervention); follow-up (T2; 12 months after intervention finished)
  N-back. It consists of indicating when the current stimulus matches the one from n steps earlier in the sequence. The load factor n can be adjusted (0-1-2-3). Correct responses : number of correct responses to targets. Omissions: number of failures to respond to targets. Comissions: number of incorrect responses to non-targets. Mean Reaction Time: mean response speed of correct responses for the whole administration.
Change from baseline cognitive flexibility at 8 weeks and at 12 months | Baseline (T0; 1 week before intervention); postraining (T1; 1 week after intervention); follow-up (T2; 12 months after intervention finished)
  Children Color Trail Test - II. Total expended time.
Change from baseline set-shifting at 8 weeks and at 12 months | Baseline (T0; 1 week before intervention); postraining (T1; 1 week after intervention); follow-up (T2; 12 months after intervention finished)
  Shifting (Five Digits Test). Total expended time.
Change from baseline attentional inhibition at 8 weeks and at 12 months | Baseline (T0; 1 week before intervention); postest (T1; 1 week after intervention); follow-up (T2; 12 months after intervention finished)
  Choosing (Five Digits Test). Total expended time.
Change from baseline behavioral inhibition at 8 weeks and at 12 months | Baseline (T0; 1 week before intervention); postest (T1; 1 week after intervention); follow-up (T2; 12 months after intervention finished)
  Go/No Go: it requires to perform an action given a letter stimuli ("p"- Go) and inhibit that action under a different set of stimuli ("r"- No-Go). After several trials the instructions are reversed ("r"-Go; "p"- No Go).
Change from baseline planning/reasoning at 8 weeks and at 12 months | Baseline (T0; 1 week before intervention); postraining (T1; 1 week after intervention); follow-up (T2; 12 months after intervention finished)
  Tower of London consists of two boards with pegs and several beads with different colors. The examiner uses the beads and the boards to present the examinee with problem-solving tasks.
Change from baseline neuroimaging (T1-weighted 3D sequence) at 8 weeks and at 12 months | Baseline (T0; 1 week before intervention); postraining (T1; 1 week after intervention); follow-up (T2; 12 months after intervention finished)
  MPRAGE sequence: TR=2300 ms, TE=2.98 ms, TI 900 ms, 240 slices, FOV=256 mm; matrix size=256x256; 1 mm isotropic voxel
Change from baseline neuroimaging (T2-weighted 3D sequence) at 8 weeks and at 12 months | Baseline (T0; 1 week before intervention); postraining (T1; 1 week after intervention); follow-up (T2; 12 months after intervention finished)
  TR=3200 ms, TE=298 ms, 256 slices, FOV=224 mm; matrix size=256x256; 0.9 mm isotropic voxel
Change from baseline neuroimaging (Diffusion Tensor Imaging sequence) at 8 weeks and at 12 months | Baseline (T0; 1 week before intervention); postraining (T1; 1 week after intervention); follow-up (T2; 12 months after intervention finished)
  Singleshot diffusion weighted EPI sequence, two adquisitions AP and PA: b=1000mm2/s, 30 directions, TR=7700 ms, TE=89 ms, flip angle 90o, slice thickness=2 mm, 1.97 mm in-plane resolution
Change from baseline neuroimaging (resting-state fMRI sequence) at 8 weeks and at 12 months | Baseline (T0; 1 week before intervention); postraining (T1; 1 week after intervention); follow-up (T2; 12 months after intervention finished)
  gradient-echo echo-planar imaging-EPI sequence: 200 volumes of 40 axial slices, TR=2500ms; TE=28ms; matrix=80x80; field of view=24cm; slice thickness=3mm; 15% interslice gap; flip angle= 80o
Change from baseline neuroimaging (clinical sequences) at 8 weeks and at 12 months | Baseline (T0; 1 week before intervention); postraining (T1; 1 week after intervention); follow-up (T2; 12 months after intervention finished)
  clinical T2 (TR/TE=5150/99 ms; 512x307 matrix, flip angle 120o, slice thickness 5 mm with a 1.5-mm interslice gap) and FLAIR sequences (TR/TE=9040/85 ms; TI= 2500; 250X171 matrix, flip angle 150o, slice thickness 5 mm)
Food-choices | Daily, over 6 weeks (training period)
  Photographs of participants' meals (breakfast, lunch, dinner).
Change from baseline Body Mass Index (BMI) and waist circumference at 8 weeks and at 12 months | Baseline (T0; 1 week before intervention); postraining (T1; 1 week after intervention); follow-up (T2; 12 months after intervention finished)
  Pediatric evaluation:
  Height (m) and weight (kg) measures will be collected and combined to report BMI (kg/m^2).
  Additionally, waist circumference (m) will be assessed.

SECONDARY OUTCOMES:
Change from baseline self-report quality of life at 8 weeks and at 12 months | Baseline (T0; 1 week before intervention); postraining (T1; 1 week after intervention); follow-up (T2; 12 months after intervention finished)
  Pediatric Quality of Life Inventory (parents' version and children's version). 23 items. Each item is scored from 0 to 4 (0=never; 4=almost always), yielding a total between 0 and 92. Higher scores mean worse quality of life.
Change from baseline social support and self-steem at 8 weeks and at 12 months | Baseline (T0; 1 week before intervention); postraining (T1; 1 week after intervention); follow-up (T2; 12 months after intervention finished)
  The Self-Perception Profile for Children (SPPC). 70 items. Each item is scored from 0 to 4 (0=never; 4=almost always), yielding a total between 0 and 280. Higher scores mean better social support and self-steem.
Change from baseline internalising and externalising problems at 8 weeks and at 12 months | Baseline (T0; 1 week before intervention); postraining (T1; 1 week after intervention); follow-up (T2; 12 months after intervention finished).
  Child Behavior Checklist. 113 items. Each item is scored from 0 to 2 (0=not true; 2= true very often or quite often). Higher scores mean more psychological and behavioral problems.
Change from baseline behavioral executive function at 8 weeks and at 12 months | Baseline (T0; 1 week before intervention); postraining (T1; 1 week after intervention); follow-up (T2; 12 months after intervention finished).
  Behavior Rating Inventory of Executive Function - II (Parents' version and Schools' version). 63 items. Higher scores mean more executive problems.
Activity and sleep patterns | Daily, during 6 weeks (the training period)
  Fitbit tracker. Number of steps and number of sleep hours.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Angeles Jurado Luque, PhD, Principal Investigator — Institute of Neuroscience. Department of Clinical Psychology and Psychobiology, University of Barcelona
Locations (1):
- Neuroscience Institute. Department of Clinical Psychology and Psychobiology, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sanchez-Castaneda C, Luis-Ruiz S, Ramon-Krauel M, Lerin C, Sanchez C, Miro N, Martinez S, Garolera M, Jurado MA. Executive Function Training in Childhood Obesity: Food Choice, Quality of Life, and Brain Connectivity (TOuCH): A Randomized Control Trial Protocol. Front Pediatr. 2021 Feb 24;9:551869. doi: 10.3389/fped.2021.551869. eCollection 2021. PMID 33718294